CLINICAL TRIAL: NCT01442480
Title: Cardioprotective Effects of Omega-3 Fatty Acids Supplementation in Healthy Older Subjects Exposed to Air Pollution Particles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Environmental Protection Agency (EPA) (U.S. Federal Agency)
Responsible Party: Principal Investigator, Haiyan Tong, Principal Investigator, Environmental Protection Agency (EPA)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: Omegacon
Record Dates: First submitted 2011-09-26; First posted 2011-09-28 (Estimated); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Healthy
Keywords: air pollution; fatty acid supplementation
MeSH Terms: interventions — Fish Oils; Olive Oil

STUDY DESIGN:
Who Masked: Participant, Investigator

ARMS (2):
- Fish oil (Experimental)
  Interventions: Dietary Supplement: Fish oil
- Olive oil (Experimental)
  Interventions: Dietary Supplement: Olive oil

INTERVENTIONS:
Dietary Supplement: Fish oil — Subjects (ages 50 to 75 years), were randomly assigned to receive 3 g/d of fish oil (1.2 g eicosapentaenoic acid and 0.82 g docosahexaenoic acid) for 28 d.
  Arms: Fish oil
Dietary Supplement: Olive oil — Subjects (ages 50 to 75 years) were randomly assigned to receive 3 g/d of olive oil for 28 d.
  Arms: Olive oil

SUMMARY:
Exposure to ambient levels of air pollution increases cardiovascular morbidity and mortality. Advanced age is among the factors associated with susceptibility to the adverse effects of air pollution. Dietary fatty acid supplementation has been shown to decrease cardiovascular risk through multiple mechanisms. This study evaluated the efficacy of supplementation with marine fish oil or olive oil in protecting against cardiovascular effects induced by controlled exposure of middle-aged healthy volunteers to concentrated ambient air pollution particles. Subjects (ages 50 to72 years), were randomly assigned to receive 3 g/d of fish oil (1.2 g eicosapentaenoic acid and 0.82 g docosahexaenoic acid), or olive oil (3g/d) for 28 d. Subjects were then exposed to concentrated ambient air pollution particles or filtered air for 2 hr on sequential days. Heart rate variability (HRV), plasma lipids, coagulation markers, and endothelial function measured by flow-mediated dilation of the brachial artery (FMD) were assessed pre-, immediately post-, and 20 hr post-exposure.

ELIGIBILITY:
Inclusion Criteria:

* Age 50-75 years old generally healthy male and female.
* Normal resting electrocardiogram.
* Oxygen saturation greater than 94% at the time of physical exam.

Exclusion Criteria:

* A history of angina, cardiac arrhythmias, congestive heart failure, and ischemic myocardial infarction or coronary bypass surgery.
* Cardiac pacemaker.
* Uncontrolled hypertension (> 150 systolic, > 90 diastolic).
* Neurodegenerative diseases such as Parkinson's and Alzheimer disease.
* A history of chronic illnesses such as diabetes, cancer (possible exception for history of nonmelanoma skin cancer), rheumatologic diseases, immunodeficiency state, significant chronic respiratory diseases such as chronic obstructive pulmonary disease or severe asthma.
* A history of migraine headache.
* History of bleeding diathesis.
* Currently taking beta-blockers to control hypertension and/or arrhythmias.
* Use of oral anticoagulants.
* Participants must refrain from all over-the-counter nonsteroidal anti-inflammatory drugs for a period of two weeks prior to exposure. Low-dose aspirin will be acceptable. Medications not specifically mentioned here may be reviewed by the investigators prior to a participant's inclusion in the study.
* Allergies to fish or omega-3 fatty acids.
* Subjects are on prescriptions taking omega-3 fish oil as therapy.
* Subjects will be required to avoid taking omega-3 fatty acids or having more than one 4-6 oz/serving of all types of fish and shellfish, walnuts, flaxseeds and flaxseed oil, rapeseed oil, canola oil, soybeans and soy products, omega-3 fortified eggs, and cod liver oil for two weeks before and during the study.
* Subjects will be required to avoid taking antioxidants (e.g., beta-carotene, selenium, vitamin C, vitamin E, zinc) for two weeks before and during the study.
* Subjects will be required to use olive oil exclusively for cooking, dressings, and sauces during the study and to avoid other vegetable oils because of their omega-3 contents.
* Because of reported cardioprotective effects of red wine, subjects will be required to avoid drinking red wine during the study.
* Subjects who are currently smoking or have smoking history within 1 year of study (defined as more than one pack of cigarettes in the past year) or have a greater than/equal to a 5 pack year smoking history.
* No exposure will be conducted within 2 weeks of a respiratory tract infection.
* Subject is pregnant, attempting to become pregnant or breastfeeding.
* Unspecified illnesses, which in the judgment of the investigators might increase the risk associated with PM inhalation will be a basis for exclusion.
* Have an allergy to latex.
* History of skin allergy to tape or electrodes.

Ages: 50 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2009-06; Primary Completion 2010-08 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Heart rate variability changes | pre-, immediately post-, and 20 hr post-air pollution exposure

SECONDARY OUTCOMES:
endothelial function changes measured by flow-mediated dilation of the brachial artery | pre-, immediately post-, and 20 hr post-air pollution exposure

CONTACTS AND LOCATIONS:
Locations (1):
- EPA Human Studies Facility, Chapel Hill, North Carolina, United States